CLINICAL TRIAL: NCT02688036
Title: Phase III Randomized Study of Hypofractionated vs Conventionally Fractionated Concurrent Chemo-radiotherapy for Limited Disease Small Cell Lung Cancer
Brief Title: Hypofractionated vs. Conventionally Fractionated Concurrent CRT for LD-SCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Sun Yat-sen University (Other); Fudan University (Other); West China Hospital (Other); Zhejiang Cancer Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Luhua Wang, Vice President of Cancer hospital of CAMS, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-L-045/2
Record Dates: First submitted 2015-11-20; First posted 2016-02-23 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Carcinoma, Small Cell; Lung Neoplasms
Keywords: Limited Disease Small Cell Lung Cancer; concurrent chemoradiotherapy; dose fractionation
MeSH Terms: conditions — Carcinoma, Small Cell; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hypofractionated CRT (Experimental): hypofractionated concurrent chemoradiotherapy
  Interventions: Radiation: hypofractionated concurrent chemoradiotherapy
- conventionally fractionated CRT (Active Comparator): conventionally fractionated concurrent chemoradiotherapy
  Interventions: Radiation: conventionally fractionated concurrent chemoradiotherapy

INTERVENTIONS:
Radiation: hypofractionated concurrent chemoradiotherapy — For patients with Limited Disease Small Cell Lung Cancer, 45Gy/15F of radiotherapy with concurrent chemotherapy will be used in experimental arm.
  Arms: hypofractionated CRT
Radiation: conventionally fractionated concurrent chemoradiotherapy — For patients with Limited Disease Small Cell Lung Cancer, 60Gy/30F of radiotherapy with concurrent chemotherapy will be used in the control arm.
  Arms: conventionally fractionated CRT

SUMMARY:
The purpose of this study is to determine whether hypofractionated concurrent chemo-radiotherapy has the same efficiency as conventionally fractionated concurrent chemo-radiotherapy in Limited Disease Small Cell Lung Cancer.

DETAILED DESCRIPTION:
For patients with Limited Disease Small Cell Lung Cancer, 45Gy/15F of radiotherapy with concurrent chemotherapy will be used in experimental arm. While 60Gy/30F of radiotherapy with concurrent chemotherapy will be used in the control arm. Both survival and toxicity of the two arms will be observed and compared.

ELIGIBILITY:
Inclusion Criteria:

* 18~70 years old, ECOG 0-2
* patients with histologically or cytologically proved small cell lung cancer
* Limited disease (LD), was characterized by tumors confined to one hemithorax. It may include ipsilateral hilar, both mediastinum and both supraclavicular nodes. Metastatic lymph nodes were defined as lymph nodes with short diameter of more than 1cm or FDG uptake in PET. The thickness of pleural effusion was less than 1cm unless malignant pleural effusion was cytologically proved. In a word, stage I-IIIB excluding the patients with lung metastases should be defined as LD according to AJCC cancer staging 7th edition.
* No progression after 2 cycles of chemotherapy with EP.
* No prior history of anti-tumor treatment.
* No severe internal diseases and no organ dysfunction
* Written informed consent provided and

Exclusion Criteria:

* Malignant tumors of other sites. Non melanoma skin cancer and Cervical carcinoma in situ were not included if curable.
* Active heart disease or acute myocardial infarction happen in six months.
* Psychiatric history.
* Pregnant woman or woman need to breast feed or woman with positive chorionic gonadotrophin (HCG)
* Uncontrolled diabetes or hypertension
* Interstitial pneumonia or Active pulmonary fibrosis
* Acute bacterial or fungal infection
* Oral or intravenous use of steroids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2 years

SECONDARY OUTCOMES:
disease free survival | 2 years
local-regional failure (Incidence of tumor recurrence in local or regional area) | 2 years
  Incidence of tumor recurrence in local or regional area
toxicity (Incidence of radiotherapy and chemotherapy induced toxicities assessed by CTCAE v 4.0) | 2 year
  Incidence of radiotherapy and chemotherapy induced toxicities assessed by CTCAE v 4.0

CONTACTS AND LOCATIONS:
Overall Officials: LuHua Wang, MD, Principal Investigator — Cancer Hospital of CAMS
Locations (1):
- Cancer Insititute and Hosiptal of Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Govindan R, Page N, Morgensztern D, Read W, Tierney R, Vlahiotis A, Spitznagel EL, Piccirillo J. Changing epidemiology of small-cell lung cancer in the United States over the last 30 years: analysis of the surveillance, epidemiologic, and end results database. J Clin Oncol. 2006 Oct 1;24(28):4539-44. doi: 10.1200/JCO.2005.04.4859. PMID 17008692
- [Background] Pignon JP, Arriagada R, Ihde DC, Johnson DH, Perry MC, Souhami RL, Brodin O, Joss RA, Kies MS, Lebeau B, et al. A meta-analysis of thoracic radiotherapy for small-cell lung cancer. N Engl J Med. 1992 Dec 3;327(23):1618-24. doi: 10.1056/NEJM199212033272302. PMID 1331787
- [Background] Warde P, Payne D. Does thoracic irradiation improve survival and local control in limited-stage small-cell carcinoma of the lung? A meta-analysis. J Clin Oncol. 1992 Jun;10(6):890-5. doi: 10.1200/JCO.1992.10.6.890. PMID 1316951
- [Background] Murray N, Coy P, Pater JL, Hodson I, Arnold A, Zee BC, Payne D, Kostashuk EC, Evans WK, Dixon P, et al. Importance of timing for thoracic irradiation in the combined modality treatment of limited-stage small-cell lung cancer. The National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 1993 Feb;11(2):336-44. doi: 10.1200/JCO.1993.11.2.336. PMID 8381164
- [Background] Jeremic B, Shibamoto Y, Acimovic L, Milisavljevic S. Initial versus delayed accelerated hyperfractionated radiation therapy and concurrent chemotherapy in limited small-cell lung cancer: a randomized study. J Clin Oncol. 1997 Mar;15(3):893-900. doi: 10.1200/JCO.1997.15.3.893. PMID 9060525
- [Background] Takada M, Fukuoka M, Kawahara M, Sugiura T, Yokoyama A, Yokota S, Nishiwaki Y, Watanabe K, Noda K, Tamura T, Fukuda H, Saijo N. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with cisplatin and etoposide for limited-stage small-cell lung cancer: results of the Japan Clinical Oncology Group Study 9104. J Clin Oncol. 2002 Jul 15;20(14):3054-60. doi: 10.1200/JCO.2002.12.071. PMID 12118018
- [Background] Kubota K, Hida T, Ishikura S, Mizusawa J, Nishio M, Kawahara M, Yokoyama A, Imamura F, Takeda K, Negoro S, Harada M, Okamoto H, Yamamoto N, Shinkai T, Sakai H, Matsui K, Nakagawa K, Shibata T, Saijo N, Tamura T; Japan Clinical Oncology Group. Etoposide and cisplatin versus irinotecan and cisplatin in patients with limited-stage small-cell lung cancer treated with etoposide and cisplatin plus concurrent accelerated hyperfractionated thoracic radiotherapy (JCOG0202): a randomised phase 3 study. Lancet Oncol. 2014 Jan;15(1):106-13. doi: 10.1016/S1470-2045(13)70511-4. Epub 2013 Dec 3. PMID 24309370
- [Background] Auperin A, Arriagada R, Pignon JP, Le Pechoux C, Gregor A, Stephens RJ, Kristjansen PE, Johnson BE, Ueoka H, Wagner H, Aisner J. Prophylactic cranial irradiation for patients with small-cell lung cancer in complete remission. Prophylactic Cranial Irradiation Overview Collaborative Group. N Engl J Med. 1999 Aug 12;341(7):476-84. doi: 10.1056/NEJM199908123410703. PMID 10441603
- [Background] Carney DN, Mitchell JB, Kinsella TJ. In vitro radiation and chemotherapy sensitivity of established cell lines of human small cell lung cancer and its large cell morphological variants. Cancer Res. 1983 Jun;43(6):2806-11. PMID 6303568
- [Background] Turrisi AT 3rd, Kim K, Blum R, Sause WT, Livingston RB, Komaki R, Wagner H, Aisner S, Johnson DH. Twice-daily compared with once-daily thoracic radiotherapy in limited small-cell lung cancer treated concurrently with cisplatin and etoposide. N Engl J Med. 1999 Jan 28;340(4):265-71. doi: 10.1056/NEJM199901283400403. PMID 9920950
- [Background] Movsas B, Moughan J, Komaki R, Choy H, Byhardt R, Langer C, Goldberg M, Graham M, Ettinger D, Johnstone D, Abrams R, Munden R, Starkschall G, Owen J. Radiotherapy patterns of care study in lung carcinoma. J Clin Oncol. 2003 Dec 15;21(24):4553-9. doi: 10.1200/JCO.2003.04.018. Epub 2003 Nov 3. PMID 14597743
- [Background] Salama JK, Hodgson L, Pang H, Urbanic JJ, Blackstock AW, Schild SE, Crawford J, Bogart JA, Vokes EE; Cancer and Leukemia Group B. A pooled analysis of limited-stage small-cell lung cancer patients treated with induction chemotherapy followed by concurrent platinum-based chemotherapy and 70 Gy daily radiotherapy: CALGB 30904. J Thorac Oncol. 2013 Aug;8(8):1043-9. doi: 10.1097/JTO.0b013e318293d8a4. PMID 23715301
- [Background] Gazula A, Baldini EH, Chen A, Kozono D. Comparison of once and twice daily radiotherapy for limited stage small-cell lung cancer. Lung. 2014 Feb;192(1):151-8. doi: 10.1007/s00408-013-9518-9. Epub 2013 Oct 27. PMID 24162870
- [Background] Withers HR, Taylor JM, Maciejewski B. The hazard of accelerated tumor clonogen repopulation during radiotherapy. Acta Oncol. 1988;27(2):131-46. doi: 10.3109/02841868809090333. PMID 3390344
- [Background] Spiro SG, James LE, Rudd RM, Trask CW, Tobias JS, Snee M, Gilligan D, Murray PA, Ruiz de Elvira MC, O'Donnell KM, Gower NH, Harper PG, Hackshaw AK; London Lung Cancer Group. Early compared with late radiotherapy in combined modality treatment for limited disease small-cell lung cancer: a London Lung Cancer Group multicenter randomized clinical trial and meta-analysis. J Clin Oncol. 2006 Aug 20;24(24):3823-30. doi: 10.1200/JCO.2005.05.3181. PMID 16921033
- [Background] Liu HH, Wang X, Dong L, Wu Q, Liao Z, Stevens CW, Guerrero TM, Komaki R, Cox JD, Mohan R. Feasibility of sparing lung and other thoracic structures with intensity-modulated radiotherapy for non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2004 Mar 15;58(4):1268-79. doi: 10.1016/j.ijrobp.2003.09.085. PMID 15001272
- [Background] Chang JY, Dong L, Liu H, Starkschall G, Balter P, Mohan R, Liao Z, Cox JD, Komaki R. Image-guided radiation therapy for non-small cell lung cancer. J Thorac Oncol. 2008 Feb;3(2):177-86. doi: 10.1097/JTO.0b013e3181622bdd. PMID 18303441
- [Background] Xia B, Chen GY, Cai XW, Zhao JD, Yang HJ, Fan M, Zhao KL, Fu XL. Is involved-field radiotherapy based on CT safe for patients with limited-stage small-cell lung cancer? Radiother Oncol. 2012 Feb;102(2):258-62. doi: 10.1016/j.radonc.2011.10.003. Epub 2011 Nov 5. PMID 22056536
- [Background] Xia B, Hong LZ, Cai XW, Zhu ZF, Liu Q, Zhao KL, Fan M, Mao JF, Yang HJ, Wu KL, Fu XL. Phase 2 study of accelerated hypofractionated thoracic radiation therapy and concurrent chemotherapy in patients with limited-stage small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2015 Mar 1;91(3):517-23. doi: 10.1016/j.ijrobp.2014.09.042. Epub 2014 Dec 3. PMID 25481679
- [Background] Giuliani ME, Lindsay PE, Sun A, Bezjak A, Le LW, Brade A, Cho J, Leighl NB, Shepherd FA, Hope AJ. Locoregional failures following thoracic irradiation in patients with limited-stage small cell lung carcinoma. Radiother Oncol. 2012 Feb;102(2):263-7. doi: 10.1016/j.radonc.2011.12.009. Epub 2012 Jan 28. PMID 22285072
- [Background] Socha J, Guzowska A, Tyc-Szczepaniak D, Szczesna A, Kepka L. Hypofractionated conformal radiotherapy in combination with chemotherapy in limited disease small cell lung cancer patients. Pneumonol Alergol Pol. 2014;82(2):105-15. doi: 10.5603/PiAP.2014.0016. PMID 24615194
- [Background] Padda SK, Burt BM, Trakul N, Wakelee HA. Early-stage non-small cell lung cancer: surgery, stereotactic radiosurgery, and individualized adjuvant therapy. Semin Oncol. 2014 Feb;41(1):40-56. doi: 10.1053/j.seminoncol.2013.12.011. Epub 2013 Dec 12. PMID 24565580
- [Background] Cannon DM, Mehta MP, Adkison JB, Khuntia D, Traynor AM, Tome WA, Chappell RJ, Tolakanahalli R, Mohindra P, Bentzen SM, Cannon GM. Dose-limiting toxicity after hypofractionated dose-escalated radiotherapy in non-small-cell lung cancer. J Clin Oncol. 2013 Dec 1;31(34):4343-8. doi: 10.1200/JCO.2013.51.5353. Epub 2013 Oct 21. PMID 24145340
- [Background] Din OS, Harden SV, Hudson E, Mohammed N, Pemberton LS, Lester JF, Biswas D, Magee L, Tufail A, Carruthers R, Sheikh G, Gilligan D, Hatton MQ. Accelerated hypo-fractionated radiotherapy for non small cell lung cancer: results from 4 UK centres. Radiother Oncol. 2013 Oct;109(1):8-12. doi: 10.1016/j.radonc.2013.07.014. Epub 2013 Oct 3. PMID 24094626
- [Background] Osti MF, Agolli L, Valeriani M, Falco T, Bracci S, De Sanctis V, Enrici RM. Image guided hypofractionated 3-dimensional radiation therapy in patients with inoperable advanced stage non-small cell lung cancer. Int J Radiat Oncol Biol Phys. 2013 Mar 1;85(3):e157-63. doi: 10.1016/j.ijrobp.2012.10.012. Epub 2012 Nov 20. PMID 23182393
- [Background] Amini A, Lin SH, Wei C, Allen P, Cox JD, Komaki R. Accelerated hypofractionated radiation therapy compared to conventionally fractionated radiation therapy for the treatment of inoperable non-small cell lung cancer. Radiat Oncol. 2012 Mar 15;7:33. doi: 10.1186/1748-717X-7-33. PMID 22420631
- [Background] Kwint M, Uyterlinde W, Nijkamp J, Chen C, de Bois J, Sonke JJ, van den Heuvel M, Knegjens J, van Herk M, Belderbos J. Acute esophagus toxicity in lung cancer patients after intensity modulated radiation therapy and concurrent chemotherapy. Int J Radiat Oncol Biol Phys. 2012 Oct 1;84(2):e223-8. doi: 10.1016/j.ijrobp.2012.03.027. Epub 2012 May 5. PMID 22560551
- [Background] Palma DA, Senan S, Oberije C, Belderbos J, de Dios NR, Bradley JD, Barriger RB, Moreno-Jimenez M, Kim TH, Ramella S, Everitt S, Rengan R, Marks LB, De Ruyck K, Warner A, Rodrigues G. Predicting esophagitis after chemoradiation therapy for non-small cell lung cancer: an individual patient data meta-analysis. Int J Radiat Oncol Biol Phys. 2013 Nov 15;87(4):690-6. doi: 10.1016/j.ijrobp.2013.07.029. Epub 2013 Sep 10. PMID 24035329
- [Background] Stephans KL, Djemil T, Diaconu C, Reddy CA, Xia P, Woody NM, Greskovich J, Makkar V, Videtic GM. Esophageal dose tolerance to hypofractionated stereotactic body radiation therapy: risk factors for late toxicity. Int J Radiat Oncol Biol Phys. 2014 Sep 1;90(1):197-202. doi: 10.1016/j.ijrobp.2014.05.011. Epub 2014 Jul 8. PMID 25015204
- [Background] Palma DA, Senan S, Tsujino K, Barriger RB, Rengan R, Moreno M, Bradley JD, Kim TH, Ramella S, Marks LB, De Petris L, Stitt L, Rodrigues G. Predicting radiation pneumonitis after chemoradiation therapy for lung cancer: an international individual patient data meta-analysis. Int J Radiat Oncol Biol Phys. 2013 Feb 1;85(2):444-50. doi: 10.1016/j.ijrobp.2012.04.043. Epub 2012 Jun 9. PMID 22682812
- [Background] De Ruysscher D, Bremer RH, Koppe F, Wanders S, van Haren E, Hochstenbag M, Geeraedts W, Pitz C, Simons J, ten Velde G, Dohmen J, Snoep G, Boersma L, Verschueren T, van Baardwijk A, Dehing C, Pijls M, Minken A, Lambin P. Omission of elective node irradiation on basis of CT-scans in patients with limited disease small cell lung cancer: a phase II trial. Radiother Oncol. 2006 Sep;80(3):307-12. doi: 10.1016/j.radonc.2006.07.029. Epub 2006 Sep 1. PMID 16949169
- [Background] Colaco R, Sheikh H, Lorigan P, Blackhall F, Hulse P, Califano R, Ashcroft L, Taylor P, Thatcher N, Faivre-Finn C. Omitting elective nodal irradiation during thoracic irradiation in limited-stage small cell lung cancer--evidence from a phase II trial. Lung Cancer. 2012 Apr;76(1):72-7. doi: 10.1016/j.lungcan.2011.09.015. Epub 2011 Oct 19. PMID 22014897
- [Background] van Loon J, De Ruysscher D, Wanders R, Boersma L, Simons J, Oellers M, Dingemans AM, Hochstenbag M, Bootsma G, Geraedts W, Pitz C, Teule J, Rhami A, Thimister W, Snoep G, Dehing-Oberije C, Lambin P. Selective nodal irradiation on basis of (18)FDG-PET scans in limited-disease small-cell lung cancer: a prospective study. Int J Radiat Oncol Biol Phys. 2010 Jun 1;77(2):329-36. doi: 10.1016/j.ijrobp.2009.04.075. Epub 2009 Sep 24. PMID 19782478
- [Background] Shirvani SM, Komaki R, Heymach JV, Fossella FV, Chang JY. Positron emission tomography/computed tomography-guided intensity-modulated radiotherapy for limited-stage small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):e91-7. doi: 10.1016/j.ijrobp.2010.12.072. Epub 2011 Apr 12. PMID 21489716